CLINICAL TRIAL: NCT05889598
Title: Effects of a Resistance Exercise Programme on Risk of Osteoporosis and Osteoarthritis in Females
Brief Title: Resistance Exercise Training to Improve Bone and Articular Cartilage Health in Women
Acronym: REPROOF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Loughborough University (Other)
Collaborators: Versus Arthritis (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Senior Lecturer in Human Biology, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 304156
Record Dates: First submitted 2022-04-26; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Osteoporosis; Osteoarthritis
Keywords: Exercise; Explosive high-velocity; Bone mineral density; Knee joint; Neuromuscular; Biomarkers
MeSH Terms: conditions — Osteoporosis; Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ballistic resistance exercise training (Experimental): This arm will perform the exercises in a hack squat machine using low loads and explosive high-velocity (as if trying to jump)
  Interventions: Other: Ballistic Resistance Lower Body Strength Training
- Conventional resistance exercise training (Experimental): This arm will perform the exercises in a hack squat machine using high-load and low-velocity (conventional training)
  Interventions: Other: Conventional Resistance Lower Body Strength Training
- Control (No Intervention): Continue usual life

INTERVENTIONS:
Other: Ballistic Resistance Lower Body Strength Training — The exercise programme involves two supervised sessions per week at University. Each session will involve 30-40 minutes of exercise, comprising warm-up , two main exercises: a hack squat and calf raise using a hack squat machine, and core exercises. After a warm-up period involving 5 minutes cycling and one set of 5 conventional repetitions at 40%1RM, the ballistic training group will complete eccentric phase hack squat exercise in approximately 3 seconds and the concentric phase as fast as possible with throwing type contractions. If participants can, participants will be allowed to take off in the concentric phase. To maintain high velocity in this group, lower loads will be used compared to the conventional group. The load will be decided according to regular maximal muscular strength test (1RM) to use of the correct weight for training (in proportion to the strength). Participants will start off using light weights and these will increase as participants become stronger.
  Arms: Ballistic resistance exercise training
Other: Conventional Resistance Lower Body Strength Training — The exercise programme involves two supervised sessions per week at Loughborough University. Each session will involve 30-40 minutes of exercise, comprising warm-up , two main exercises: a hack squat and calf raise using a hack squat machine, and core exercises. After a warm-up period involving 5 minutes cycling and one set of 5 conventional repetitions at 40% of 1RM, the conventional training group will complete eccentric and concentric phases of hack squatting exercises for approximately 3 seconds each, with appropriate breathing techniques. The load will be decided according to regular maximal muscular strength test (1RM) to use of the correct weight for training (in proportion to the strength). Participants will start off using light weights and these will increase as participants become stronger.
  Arms: Conventional resistance exercise training

SUMMARY:
Osteoarthritis (degenerative joint disease) and osteoporosis (weak and fragile bones) are common conditions, particularly in women after menopause, and become even more common as we get older. Aging is also associated with sarcopenia, the progressive loss of muscle strength and mass with age. In this three-arm study, the effect of resistance exercise programs with different parameters (such as velocity and load) on various outcomes, including structural changes (bone mineral density, cartilage composition, muscle size), physical function, and biomarkers will be compared.

DETAILED DESCRIPTION:
Resistance exercise is effective in improving several risk factors for osteoporosis and osteoarthritis, and is recommended to prevent and manage both conditions, and is also known to counteract sarcopenia. Overall, there is little and inconsistent evidence on the effects of exercise parameters (such as velocity) for the prevention of osteoporosis and osteoarthritis, neither is there a comparison of different velocities on structural parameters and biomarkers. Although osteoporosis and osteoarthritis take a long time to develop, it is possible to look at changes in risk using scans of bones and joints -Dual-Energy X-ray absorptiometry (DXA), peripheral Quantitative Computed Tomography (pQCT), and Magnetic Resonance Imaging (MRI)-, blood and/or urine samples and symptoms.

This study aims to examine the effect of two different resistance exercise interventions (explosive high-velocity vs high-load low-velocity training) on structural changes on bone, articular knee and/or hip cartilage and muscle, as well as biomarkers.

The study will be a 32-week long randomized controlled trial including two exercise groups and one non-exercising control group.

Screening and baseline measurements will then be taken when anonymization is completed. Once participants have completed baseline testing, participants will be randomly assigned to one of the exercise groups or control groups using a block randomization technique. Participants will choose an envelope, prepared in batches of 11, which will contain a note saying either 'ballistic' or 'conventional or 'control' with a ratio of 4:4:3. This is to allow for greater drop-out in the exercise groups. It is not possible to blind the participant or researchers supervising the intervention to the group allocation.

The required exercise program involves two supervised sessions per week at Loughborough University, each lasting no longer than 60 minutes per session. Each session will involve 30-40 minutes of exercise and time to check any symptoms or queries with participants.

The exercises are designed to strengthen major muscle groups of the trunk and lower body, as well as to load bones that are affected by osteoporosis and the knee and hip joints that are commonly affected by osteoarthritis. Each exercise training session will take 30-40 minutes and include some whole-body warm-up and trunk exercises before completing the two main exercises: a hack squat and calf raise. These two main exercises will be done using resistance (weight training) machines in a dedicated exercise facility. Investigators chose a hack squat machine as it exercises many muscle groups and skeletal sites in one exercise, including the spine and lower limb rather than a small area. Additionally, it supports the spine, making it safe and comfortable to use.

The intervention will be personalized to the individual's ability, and loads will steadily increase as the participant improves. The load will be decided according to maximal muscular strength determined by calculation of 1-repetition maximum which will be renewed every month to monitor the progress of their muscle strength and use of the correct weight for training (in proportion to the strength). Participants will start off using light weights and these will increase as participants become stronger.

The two exercise groups will follow the same exercise programmes but using different speeds and weights: The conventional training group will perform the exercises slowly (conventionally), whilst the ballistic group will use lower loads and higher velocity as if trying to jump. Participants will be carefully guided and coached to perform all the exercises correctly and all the exercise training sessions will be supervised by qualified researchers to ensure safety throughout the study.

The control group will be asked to maintain their usual exercise and diet. Follow-up measurements will take place 16 and 32 weeks after the commencement of the exercise programme.

The sample size calculation is based on detecting differences in bone mineral density between each exercise group and the control group. Using an effect size of 0.75 (considered clinically meaningful), alpha of 0.05, and beta errors of 0.95, approximately 28 participants are needed for each group. However, the final sample size should cover a possible number of withdrawals. To allow for a 30% drop-out rate in exercise groups, 110 participants will be recruited for the study.

All data will be reported in the final work; any missing data will be accounted for with reasons for it missing. All measures described in the methodology will be reported, whether results are statistically significant or not. Data from all eligible participants will be included in an intention-to-treat analysis. Multiple imputation will be used for addressing the presence of missing data. The analysis will be repeated in good adherers i.e. those who attended at least 90% of the exercise sessions.

Descriptive statistics will be calculated to give information on mean values and variation (standard deviation) of the cohort. Normal distribution will be analysed using Shapiro-Wilk test. If variance is shown to be homogenous and distribution normal within the population then repeated measures analysis of variance (RM-ANOVA) will detect any significant differences between group (exercise versus control), time (baseline versus post-intervention) or group x time interaction.

ELIGIBILITY:
Inclusion Criteria:

* Women between 50-70 years;
* Experienced last menstrual cycle, hormonal contraception or menopausal hormone replacement therapy at least five years ago;
* Independent living and able to come into the university;
* Healthy women: not previously diagnosed with osteoporosis or knee osteoarthritis, other major medical conditions;
* Able to understand English.

Exclusion Criteria:

* Any existing symptomatic knee, hip, back injury or any medical conditions or injuries which would affect the ability or safety to perform exercise or influence bone/cartilage, including unstable angina, uncontrolled hypertension, a history of heart failure, and a history of cardiovascular disease and conditions;
* Taking medication affecting bone/cartilage metabolism;
* Regular (>once per week on average) participation in resistance training with loading greater than bodyweight or in high impact (impact greater than jogging);
* Blood pressure exceeding 150/90 mmHg;
* BMI > 30 kg/m2;
* Contraindications to MRI or DXA (e.g. Metallic implants);
* Osteoporotic (FRAX score according to which the participant would be advised to seek treatment);
* Fracture within the past year.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Femoral neck bone mineral content from baseline | 32nd week
  (g) measured by DXA
Change in Femoral neck bone mineral density from baseline | 32nd week
  (g/cm^2) measured by DXA

SECONDARY OUTCOMES:
Bone Mineral Content (Femur) | Baseline, 16th and 32nd weeks
  Proximal Femur bone will be assessed in "g" by DXA
Bone Mineral Density (Femur) | Baseline, 16th and 32nd weeks
  Proximal femur bone will be assessed (g/cm^2) by DXA
Bone Mineral Content (Spine) | Baseline, 16th and 32nd weeks
  Lumbar spine bone will be assessed (g) by DXA
Bone Mineral Density (Spine) | Baseline, 16th and 32nd weeks
  Lumbar spine will be assessed (g/cm^2) by DXA
bone mineral content (Forearm) | Baseline, 16th and 32nd weeks
  Forearm bone will be assessed (g) by DXA
bone mineral density (Forearm) | Baseline, 16th and 32nd weeks
  Forearm bone will be assessed (g/cm^2) by DXA
Bone mineral content (Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone will be assessed (g) by DXA
bone mineral density (Lower Leg) | Baseline, 16th and 32nd weeks
  Tibia bone will be assessed (g/cm^2) by DXA
Bone mineral content (Total body) | Baseline, 16th and 32nd weeks
  Whole body will be assessed (g) by DXA
bone mineral density (Total Body) | Baseline, 16th and 32nd weeks
  Whole body will be assessed (g/cm^2) by DXA
cortical bone subdensity (Forearm) | Baseline, 16th and 32nd weeks
  Radius bone 4% (mg/cm^3) measured by pQCT
total bone density (Forearm) | Baseline, 16th and 32nd weeks
  Radius bone 4% (mg/cm^3) measured by pQCT
trabecular bone density (Forearm) | Baseline, 16th and 32nd weeks
  Radius bone 4% (mg/cm^3) measured by pQCT
bone total density (Forearm) | Baseline, 16th and 32nd weeks
  Radius bone 66% (mg/cm^3) measured by pQCT
cortical bone density (Forearm) | Baseline, 16th and 32nd weeks
  Radius bone 66% (mg/cm^3) measured by pQCT
total bone density (Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone 4% (mg/cm^3) measured by pQCT
trabecular bone density (Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone 4% (mg/cm^3) measured by pQCT
cortical bone subdensity (Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone 4% (mg/cm^3) measured by pQCT
bone total density (Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone 38% (mg/cm^3) measured by pQCT
cortical bone density (Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone 38% (mg/cm^3) measured by pQCT
total bone density (66% of Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone 66% (mg/cm^3) measured by pQCT
cortical density (Lower leg) | Baseline, 16th and 32nd weeks
  Tibia bone 66% (mg/cm^3) measured by pQCT
T2 relaxation time | Baseline and 32nd week
  Knee joint cartilage (ms) measured by MRI
cartilage thickness | Baseline and 32nd week
  Knee joint cartilage (mm) measured by MRI
Change in bone turnover biomarkers (CTX-1 and P1NP) in bodily samples | Baseline, 16th and 32nd weeks
  Serum/urine will be assessed by ELISA kits
Lower limb power | Baseline, 16th and 32nd weeks
  (W) measured during Hack squat action
Lower limb force | Baseline, 16th and 32nd weeks
  (N) measured during Hack squat action
Lower limb velocity | Baseline, 16th and 32nd weeks
  (m/s) measured during Hack squat action
Quadriceps cross-sectional area | Baseline and 32nd week
  (cm^2) measured by MRI
Triceps surae cross-sectional area | Baseline and 32nd week
  (cm^2) measured by pQCT
Lower extremity functioning | Baseline, 16th and 32nd weeks
  (total score in points) using Short Physical Performance Battery. SPPB scores range from zero to 12 possible points. SPPB score of 10 or greater for persons with no mobility disability indicates robustness.
Mobility/agility | Baseline, 16th and 32nd weeks
  The timed Up and Go test is rated on a scale from 1 to 5 where 1 indicates "normal function" and 5 indicates "severely abnormal function"
Pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life following knee injury | Baseline, 16th and 32nd weeks
  the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be used for that. A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems
Pain, stiffness, and physical function of the hip and knee | Baseline, 16th and 32nd weeks
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Physical Activity Level | Baseline, 16th and 32nd weeks
  Bone-specific Physical Activity Questionnaire (BPAQ). higher scores mean higher physical and better outcomes for the study
Physical activity and inactivity level | Baseline, 16th and 32nd weeks
  International Physical Activity Questionnaire (IPAQ)
Daily calcium intake | Baseline, 16th and 32nd weeks
  (mg) Calcium Questionnaire
Static postural sway | Baseline, 16th and 32nd weeks
  anterior-posterior and medial-lateral mean velocity (cm/s) of the centre of pressure
Static postural sway (elliptical area) | Baseline, 16th and 32nd weeks
  the elliptical area (cm^2) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Brooke-Wavell, PhD, Principal Investigator — Loughborough University; Jonathan Folland, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Marques EA, Caliskan O, Brooke-Wavell K, Folland J. Feasibility of ballistic vs conventional resistance training in healthy postmenopausal women: A three-arm parallel randomised controlled trial. Maturitas. 2025 May;196:108246. doi: 10.1016/j.maturitas.2025.108246. Epub 2025 Mar 13. PMID 40106971